CLINICAL TRIAL: NCT02768584
Title: Levers and Brakes to the Therapeutic Alliance Between Patients in Hospital Full-time Psychiatric and Nurses and Caregivers
Brief Title: Construction of the Therapeutic Alliance Between Inpatient Psychiatric Patients and Nurses
Acronym: ATIASP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: PHRIP 1300036N
Record Dates: First submitted 2016-03-16; First posted 2016-05-11 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-07

CONDITIONS: Psychiatric Diseases
Keywords: severe mental illness; nursing; therapeutic alliance; psychiatric diseases
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Clarify the determinants of the construction of a Therapeutic Alliance (AT) between paramedical staff (nurses and caregivers ) and adult patients in a functional unit of full-time general psychiatric Whether the quality of Therapeutic Alliance influences the continued support outpatient , after completion of full-time hospitalization.

DETAILED DESCRIPTION:
This is a prospective, observational, multicenter inpatient units Parisian full time of the Etablissement Public Health White House (spread over 4 sites).

The study seeks to collect, on the one hand the level of AT obtained at the end of hospitalization in general adult psychiatry and, secondly, to understand how this one was built.

The AT will be measured:

* Firstly by the self-administered questionnaire STAR-P, translated into French by the "translation / back-translation" method.
* Secondly through semi-structured qualitative interviews, conducted at discharge by a health care setting or a specially trained and who did not participate directly in the patient's care included. Indeed, the questionnaires allow, through scales to measure the AT quantitative way through proposals (items) presented as so, and look for associations with some predefined decisive.

However, it is difficult to explore more complex combination of mechanisms. Conducting interviews can meet this goal. An interview grid will be conducted and organized around the search for representations and affects related relational patient / nurse(s) and caregiver(s) in the context of hospital care. The interviews will be recorded and fully transcribed. A thematic analysis will be conducted to identify the objects and themes. The inclusions in this qualitative analysis will stop when reaching the saturation process. In this type of study, it is generally necessary to include thirty people to reach saturation.

Finally, semi-structured group interviews (focus group) will be conducted by co-investigators and doctoral student psychologist caregivers with the discussion topic imposed: the AT construction. They will be directed to paramedics caregivers (nurses and caregivers) are not part of the investigation team conducting research but actively involved in care. Their goal will be to harvest their representations regarding the quality of the therapeutic relationship they're trying to build with patients. A focus group will be conducted by site (4 sites), with 5 to 12 volunteers per group.

ELIGIBILITY:
Inclusion Criteria:

* adult patient (>18 years old)
* Adult psychiatric inpatients

Exclusion Criteria:

* Patients carrying perversion disorder or paranoia
* Patients trust whose legal representative refuses participation in the survey
* patients non covered by the french health system
* non consenting patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patient suffer from pyschiatric diseases except perversion disorder or paranoia
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Therapeutic Alliance score overall with self-administered questionnaire STAR-P | day 0
  AT score overall, committed to using the self-administered questionnaire STAR-P particularly suitable for "patients with severe psychiatric disorders" (Rebecca, 2007).

SECONDARY OUTCOMES:
Number of patients reviewed in outpatient psychiatric consultation | three months after hospital discharge.
AT evaluated in patients using semi-structured interviews | day 0
  AT evaluated in patients using semi-structured interviews (20-40 minutes), led with an interview grid: research of representations and affects related relational patient / nurse (s) and caregiver ( s) under hospital care.
AT evaluated in / nurse (s) and caregiver(s) | month 6
  AT evaluated in / nurse (s) and caregiver (s), through focus group: Research performances and determinants of therapeutic alliance with caregivers.
Determinants of AT studied | day 0
  socio-demographic characteristics (age, sex, socio-professional category (CSP), educational level, profession last exercised, wage level; Marital Status; Place of birth); primary psychiatric diagnosis (ICD-10); Companion diagnostics; Total number of psychiatric hospitalizations prior to the study; which stays in Difficult Patient Unit (UMD) in Free Care, in care without consent, or at the request of a representative of the state); Stay in therapeutic isolation room during hospitalization; Length of hospital stay; Supported by a referent nurse; Highlights in the treatment period and that could presuppose an impact on the quality of care
intermediate score STAR-P: score of positive collaboration | day 0
intermediate scores STAR-P: positive contribution score | day 0
intermediate scores STAR-P: uncooperative intake score of the nursing team and caregiver | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Manuel Morvillers, PhD, Principal Investigator — centre hospitalier Maison Blanche
Locations (1):
- EPS Maison Blanche, Paris, France

IPD SHARING:
Plan to Share IPD: No
At the end of the study, patient could be informed of result of the study if they wish.
  No individual result will be communicate.